CLINICAL TRIAL: NCT06387641
Title: Effects of Life Review Intervention on Meaning in Life Among Older Adults With Disabilities：a Randomised Controlled Trial
Brief Title: Effects of Life Review Intervention on Meaning in Life Among Older Adults With Disabilities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bao Huimin (Other)
Responsible Party: Sponsor-Investigator, Bao Huimin, postgraduates, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024004
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Disabilities, Psychological
Keywords: meaning in life; life review; older adults; disabilities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants received routine community health services only.
  Interventions: Behavioral: Routine community health services
- Life Review (Experimental): In addition to regular community health services，participants receive life review interventions life review intervention once a week for 6 weeks, with each session lasting45-60 minutes.
  Interventions: Behavioral: Life review; Behavioral: Routine community health services

INTERVENTIONS:
Behavioral: Life review — Life review is a process that involves a thorough examination and reflection on one's past experiences, memories, and life events. This process often involves the identification and examination of significant themes, patterns, and lessons learned throughout one's lifespan. Through life review, individuals can gain a deeper understanding of their own identity, values, and beliefs, and how these have shaped their present circumstances and future outlooks. It can serve as a tool for personal growth, self-discovery, and the promotion of a sense of meaning and purpose in life.
  Arms: Life Review
Behavioral: Routine community health services — Routine community health services refer to a comprehensive health care service system that is government-led, community-participated, and guided by superior health institutions. It focuses on grass-roots health institutions and is staffed with general practitioners as the backbone. By rationally utilizing community resources, it provides a series of comprehensive health care services to community residents. These services center on human health, target families as the unit, cover the entire community, and aim to meet the basic health service needs of community residents.
  Specifically, routine community health services include the following aspects: Health Education, Prevention and Control, Health Care Services and so on.

SUMMARY:
The goal of this interventional study is to learn if life review works to improve the sense of meaning in life in older adults with disabilities who live at home. The main questions it aims to answer are:

Does life review enhance the sense of meaning in life of participants? Does life reviews enhance the life satisfaction of participants. Does life reviews enhance the quality of life of participants?

Researchers will compare the life review program to routine community health services to see if the life review intervention program is effective in enhancing the sense of meaning in life of older adults with disabilities who live at home.

Participants will:

Take face-to-face life review interview or routine community health service every week for 6 weeks.

Take the the questionnaire survey before and after the six-week life review intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years old
* Conform to the diagnosis of disability
* Those who scored <38 points on the Chinese version of the Meaning of Life Scale (C-MLQ)
* Conscious, able to comprehend the questionnaire, and have the ability to communicate verbally
* Voluntarily participate in the study and sign the informed consent form

Exclusion Criteria:

* With cognitive impairment
* Unable to complete the questionnaire due to their physical condition
* Participated in other psychosocial interventions during the same period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Meaning in life on the Meaning in Life Questionnaire (MLQ) at Week6 | Baseline and Week6
  The MLQ is a validated self-reported instrument assessing for sense of meaning in life, with 10 items and 2 dimensions, using a 7-point Likert scale, ranging from "totally disagree" to "totally agree" on a scale of 1-7, with a total score of 10-70, with higher scores indicating a higher level of sense of meaning in life.

SECONDARY OUTCOMES:
Change from Baseline in Life satisfaction on the Life Satisfaction In-dex A (LSIA) at Week6 | Baseline and Week6
  LSIA is a validated self-reported instrument assessing for life satisfaction. This scale has a total score of 20, with higher scores indicating greater life satisfaction.
Change from Baseline in Quality of life on the 12-Item Short Form Survey (SF-12) at Week6 | Baseline and Week6
  SF-12 is a validated self-reported instrument assessing for Quality of life. A total of 12 entries covering 8 dimensions in two areas, with a higher total score representing a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Bao, Principal Investigator — School of Nursing, Hangzhou Normal University
Locations (4):
- China (4):
  - Xixi Street Community Health Service Center, Hanzhou, Zhejiang
  - Gongchenqiao Street Community Health Service Centre, Hanzhou, Zhejiang
  - Baiyang Street Wenchao Community Health Centre, Hanzhou, Zhejiang
  - School of Nursing, Hangzhou Normal University, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lan X, Xiao H, Chen Y. Life review for Chinese older adults in nursing homes: cultural acceptance and its effects. Int Psychogeriatr. 2019 Apr;31(4):527-535. doi: 10.1017/S1041610218001084. Epub 2018 Oct 2. PMID 30277193
- [Background] Lan X, Xiao H, Chen Y, Zhang X. Effects of Life Review Intervention on Life Satisfaction and Personal Meaning Among Older Adults With Frailty. J Psychosoc Nurs Ment Health Serv. 2018 Jul 1;56(7):30-36. doi: 10.3928/02793695-20180305-01. Epub 2018 Mar 16. PMID 29538790
- [Background] Zheng M, Zhang X, Xiao H. Effects of a WeChat-Based Life Review Program for Patients With Digestive System Cancer: 3-Arm Parallel Randomized Controlled Trial. J Med Internet Res. 2022 Aug 25;24(8):e36000. doi: 10.2196/36000. PMID 36006665
- [Background] Chen Y, Sun L, Xiao H, Zheng J, Lin X. Evaluation of a WeChat-based Dyadic Life Review Program for people with advanced cancer and family caregivers: A mixed-method feasibility study. Palliat Med. 2022 Mar;36(3):498-509. doi: 10.1177/02692163211066736. Epub 2022 Feb 20. PMID 35184629